CLINICAL TRIAL: NCT06558500
Title: Uterocervical and Posterior Cervical Angle Versus Cervical Length and Bishop's Score as a Predictor of Labor Induction in Term Singleton Pregnancy: a Prospective Study
Brief Title: Uterocervical Angle Versus Cervical Length as a Predictor of Labor Induction in Term Singleton Pregnancy
Status: Completed | Type: Observational
Sponsor: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayse Gizem Yildiz, Medical doctor, Specialist of gynecology and obstetrics, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Other Study IDs: 2022/113
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Labor (Obstetrics)--Complications
Keywords: Nulliparous; labor induction; posterior cervical angle; uterocervical angle; cervical length

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: delivered vaginally with successful induction of labor
  Interventions: Procedure: Uterocervical angle
- group 2: failed induction and delivered with C/S
  Interventions: Procedure: Uterocervical angle

INTERVENTIONS:
Procedure: Uterocervical angle — With the patient in the lithotomy position and empty bladder, care was taken to avoid applying pressure to the cervix with the transvaginal probe. The cervix was aligned in the midline, and the endocervical canal was visualized throughout its length.During cervical measurement, care was taken to ensure that the internal os, external os, and entire endocervical canal were visible in the same image. With the endocervical canal, external os, and internal os linearly displayed on the screen, the angle between the endocervical canal, anterior and posterior uterine segment was measured using the ultrasound's "angle measurement" feature.For the measurement of the uterocervical angle, the first line of the angle was defined along the endocervical canal used for measuring cervical length, and the second line was drawn from the internal os along the anterior uterine segment for a minimum of two centimeters. The angle between these two lines was recorded as the uterocervical angle in the form.
  Other Names: Posterior cervical angle

SUMMARY:
Induction of labor is frequently performed in all obstetric clinics. Failed IOL has been defined in many different ways.Bishop scoring, which is a traditional and subjective method, is more frequently evaluated with cervical length, which has taken its place in preterm labor, and various ultrasonographic evaluations such as Uterocervical angle (UCA), Posterior cervical angle (PCA), cervical elastography, transvulvar ultrasonography, which have recently increased in popularity, have gained importance and led us to evaluate these parameters in our clinic. The relationship between the angles between the uterus and cervix and labor has been known for some time.

DETAILED DESCRIPTION:
Induction of labor is frequently performed in all obstetric clinics for various indications, with a worldwide spectrum ranging from 1.4 to 35%. Failed IOL has been defined in many different ways. It has been defined as a dilatation of less than 4 cm despite administration of oxytocin for 12 hours±3 hours (target 200-225 MVU or 3 contractions/10 min), induction of labor with oxytocin for at least 12-18 hours (after rupture of membranes) and a latent phase lasting 24 hours or longer, primarily considering fetal and maternal well-being. In some sources, it is defined as failure to achieve regular (e.g. every 3 minutes) uterine contractions and cervical changes with artificial rupture of membranes after at least 6-8 hours of oxytocin maintenance dose. For this reason, various subjective & ultrasonographic parameters used to predict induction success are of great importance for the evaluation of the cervix. Bishop scoring, which is a traditional and subjective method, is more frequently evaluated with cervical length, which has taken its place in preterm labor, and various ultrasonographic evaluations such as Uterocervical angle (UCA), Posterior cervical angle (PCA), cervical elastography, transvulvar ultrasonography, which have recently increased in popularity, have gained importance and led us to evaluate these parameters in our clinic.

The relationship between the angles between the uterus and cervix and labor has been known for some time.

ELIGIBILITY:
Inclusion Criteria:

37 weeks and older Nulliparity Live, singular Verteks presentation Cervical opening<3 cm Bishop score<7 Patients not in active action

Exclusion Criteria:

* Presence of contraindications to vaginal delivery (pls previa, detached pls...)
* History of previous uterine surgery
* Multiple pregnancies
* Non-vertex presentation
* Uncontrolled HT Uncontrolled DM
* Fetal distress
* Macrosomic fetus Patients in active labor

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This prospective observational study was conducted at the Department of Obstetrics and Gynecology, Ankara Etlik Hospital, between June 2024 and August 2024, on 140 term pregnancies admitted for maternal or fetal reasons , planned for labor induction.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
The efficacy of uterocervical angle | 2 days
  The efficacy of uterocervical angle in predicting labor induction success in nulliparous patients at term.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Turhan ÇAĞLAR, Study Chair — Etlik Zübeyde Hanım EAH
Locations (1):
- Etlik Zubeyde Hanım Women's Health Education Hospital, Ankara, Turkey (Türkiye)